CLINICAL TRIAL: NCT04342520
Title: Anxiety Related to the Diagnosis of Alzheimer's Disease or Related Diseases
Acronym: ADIMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02620-57
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dyads Patient / caregiver — adult patient / caregiver couples, patient are 55 years of age or older and have Alzheimer's disease or a related disease

SUMMARY:
Improving the diagnosis of neurocognitive disorders is a major public health challenge. This diagnosis occurs too late in the majority of cases, or is even sometimes non-existent for some despite the presence of clinical signs and symptoms. However, the etiological diagnosis of a TNC is crucial for the patient and his family to understand the most appropriate decisions for the future, to plan the organization of his life as long as he is able to do so, to access the clinical research, to promote dialogue between patients and their caregivers. On the contrary, a late diagnosis may be responsible for the fact that the patient and his / her family are less able to benefit from certain psychosocial interventions, services and treatments.

But the diagnostic announcement is retained. One of the negative and dreaded effects of such an announcement is the negative psychological impact. Some studies show that the diagnostic announcement would worsen the level of anxiety or depressed mood and the risk of social isolation. On the other hand, other studies show that symptoms such as anxiety, psychic distress and depression remain stable, or even decrease slightly after the announcement of the diagnosis, in patients and their relatives. However, the literature is questionable because the majority of the studies are retrospective, mono-centric, and the patient numbers are low. While the first reactions of patients may be negative after the announcement, some report resignation experiences, or form of relief, because they have finally found a clinical explanation for the symptoms encountered. While doubt or diagnostic uncertainty, as well as the feeling of not knowing the truth, seem to have a more damaging psychological impact on the patient and those around him, increasing anxiety and confusion.

The primary objective is to study if the level of anxiety 2 months after the announcement of the diagnosis of Alzheimer's disease or a related disease is not superior to the level of anxiety before the announcement with patient / caregiver.

This present study aim to explore the feasibility with 14 patients.

DETAILED DESCRIPTION:
Improving the diagnosis of neurocognitive disorders is a major public health challenge. This diagnosis occurs too late in the majority of cases, or is even sometimes non-existent for some despite the presence of clinical signs and symptoms. However, the etiological diagnosis of a TNC is crucial for the patient and his family to understand the most appropriate decisions for the future, to plan the organization of his life as long as he is able to do so, to access the clinical research, to promote dialogue between patients and their caregivers. On the contrary, a late diagnosis may be responsible for the fact that the patient and his / her family are less able to benefit from certain psychosocial interventions, services and treatments.

But the diagnostic announcement is retained. One of the negative and dreaded effects of such an announcement is the negative psychological impact. Some studies show that the diagnostic announcement would worsen the level of anxiety or depressed mood and the risk of social isolation. On the other hand, other studies show that symptoms such as anxiety, psychic distress and depression remain stable, or even decrease slightly after the announcement of the diagnosis, in patients and their relatives. However, the literature is questionable because the majority of the studies are retrospective, mono-centric, and the patient numbers are low. While the first reactions of patients may be negative after the announcement, some report resignation experiences, or form of relief, because they have finally found a clinical explanation for the symptoms encountered. While doubt or diagnostic uncertainty, as well as the feeling of not knowing the truth, seem to have a more damaging psychological impact on the patient and those around him, increasing anxiety and confusion.

The primary objective is to study if the level of anxiety 2 months after the announcement of the diagnosis of Alzheimer's disease or a related disease is not superior to the level of anxiety before the announcement with patient / caregiver.

This present study aim to explore the feasibility with 14 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients :
* Man or woman 55 years and over
* Patient received for the first time in Memory Consultation and not aware of his diagnosis
* Patient with a Mini-Mental State Assessment score (MMSE) ≥ 20
* Patient accompanied by a primary caregiver
* Patient able to provide consent to participate in research

Caregiver:

* The caregiver accompanies the patient and is considered as the main caregiver during the consultation
* is able to provide consent to participate in research

Exclusion Criteria:

* Patient living in a care homes
* Patient protected by law (under legal protection, guardianship or trusteeship)
* Patient with a hearing or visual impairment that does not allow to carry out assessments in Memory Consultation
* Patient opposing research

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient / caregiver likely to participate in the study will be identified in a memory clinic as part of their regular medical course.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety (Y-B form) of the State Trait Anxiety Inventory (STAI) scale | at inclusion
  The anxiety score (Y-B form) of the State Trait Anxiety Inventory (STAI) scale, assess the level of anxiety in daily life. The range of this score is from 20 to 80.
Anxiety (Y-B form) of the State Trait Anxiety Inventory (STAI) scale | at 2 months
  The anxiety score (Y-B form) of the State Trait Anxiety Inventory (STAI) scale, assess the level of anxiety in daily life. The range of this score is from 20 to 80.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes (HCL), Lyon, France

IPD SHARING:
Plan to Share IPD: No